CLINICAL TRIAL: NCT04243746
Title: Effects of Time Restricted Feeding on Body Weight and Metabolic Syndrome Severity in the Obese Adults
Brief Title: Time Restricted Feeding to Reduce Weight and Cardiometabolic Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RCSI & UCD Malaysia Campus (Other)
Responsible Party: Principal Investigator, Dr Chean Kooi Yau, Principal investigator, senior lecturer, RCSI & UCD Malaysia Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRF168 001
Record Dates: First submitted 2020-01-19; First posted 2020-01-28 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Obesity; Metabolic Syndrome; Pre Diabetes
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Glucose Intolerance | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Feeding +Standard Malaysian Healthy Plate(QQH) (Experimental): Subjects practise time restricted feeding (TRF) in addition to the Standard Malaysian Healthy Plate (QQH).
  Interventions: Behavioral: Time Restricted Feeding
- Standard Malaysian Healthy Plate (QQH) (Active Comparator): Subjects practise the QQH dietary plan.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Time Restricted Feeding — Subjects practise TRF (2-3 meals) as an adjunct to the QQH healthy plate diet. Subjects of the intervention group can eat during the pre-determined 8-12 hours eating window, but they are only allowed to drink water and calorie-free drinks for the remaining 12-16 hours. Subjects are allowed to decide the time of their first and the last meal of the day as long as they eat within the 8-12 hour window period. However, skipping breakfast and having late dinner are discouraged.
  Arms: Time Restricted Feeding +Standard Malaysian Healthy Plate(QQH)
Behavioral: Standard Care — Subjects practice the QQH healthy plate diet as per guidelines set by the Health Ministry the guidelines.QQH refers to a normal food plate (23cm in diameter), divided into a quarter of rice (carbohydrates), a quarter of meat (protein) and a half plate of vegetables and fruits. Additionally, no calories specification is required and snacks are discouraged.
  Arms: Standard Malaysian Healthy Plate (QQH)

SUMMARY:
The obesity rate in Malaysia is higher than the average world obesity rate. Central obesity is a component of metabolic syndrome (MetS) which is also made up of dyslipidemia, impaired glucose tolerance, and hypertension. MetS is a continuum in the risk of developing cardiometabolic complication. Time Restricted Feeding (TRF) involves an extended physiological overnight fast. Researchers believe that the timing of meal intake that matches with the circadian rhythms is as important as the calories intake to prevent obesity and its complications. The investigators hypothesize that TRF is effective in weight control and improvement of metabolic severity. Subjects will be randomized into either the control group, which practices QQH dietary plan or intervention group, which practices TRF as an adjunct to QQH dietary plan.

Subjects will be followed up at week 12 and week 24 to assess adherence, efficacy and safety of TRF.

This study intends to fill a few research gaps as follows:

1. Longer study duration of 6 months.
2. This is the first study amongst the Asian population.
3. Adherence level to TRF in real life setting is measured. This information can potentially predict the intensity level of TRF that are feasible for practice in real life and also its association with the efficacy of TRF.
4. TRF is defined as eating within a≤12-hour period and fasting for at least 12 hours per day. This is the shortest fasting window studied so far.

ELIGIBILITY:
Inclusion Criteria:

1. 20-59 years of age
2. BMI 27.5kg/m2 - 39.9kg/m2
3. Smart phone users
4. Willing to lose weight
5. Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

1. Those with history of cardiovascular disease, cerebrovascular accidents, degenerative or inflammatory diseases of the nervous system; epilepsy, malignancy, gastrointestinal disorders, thyroid disorders, diabetes or medications which could have had metabolic effects.
2. Women who are pregnant or breastfeeding.
3. Those who are currently practicing any form of intermittent fasting or newly enrolled into a dietary or slimming program within the past 3 months.
4. Subjects with any medical condition, which in the investigator's judgment may be associated with increased risk to the subject or may interfere with study assessments or outcomes.
5. Those currently on medication for chronic illness.
6. Permanent night shift worker
7. Those who need to practise Ramadan fasting during the period of this study.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Body weight (kg) | baseline - 24 weeks
  Mean body weight change will be calculated.
Systolic BP (mmHg) | baseline - 24 weeks
  This is a parameter for the calculation of metabolic syndrome severity score.
Fasting blood sugar (mmol/L) | baseline - 24 weeks
  This is a parameter for the calculation of metabolic syndrome severity score.
Waist circumference (cm) | baseline - 24 weeks
  This is a parameter for the calculation of metabolic syndrome severity score.
Serum triglyceride(mmol/L) | baseline - 24 weeks
  This is a parameter for the calculation metabolic syndrome severity score.
Serum high density lipoprotein (HDL) (mmol/L) | baseline - 24 weeks
  This is a parameter for the calculation metabolic syndrome severity score.

SECONDARY OUTCOMES:
Number of fasting hours per day | baseline - 24 weeks
  For assessment of adherence
Number of days achieving TRF | baseline-24 weeks
  For assessment of adherence
Incidence of treatment-emergent adverse events [Safety ] | baseline-24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kooi Yau Chean, Principal Investigator — RCSI & UCD Malaysia Campus
Locations (1):
- Penang General Hospital, George Town, Pulau Pinang, Malaysia